CLINICAL TRIAL: NCT05825144
Title: Therapeutic Effects of Robotic Exoskeleton-Assisted Gait Re-habilitation and Predictive Factors of Significant Improvements in Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CF21277A
Record Dates: First submitted 2023-03-19; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-03

CONDITIONS: Stroke Sequelae
Keywords: robotic rehabilitation; stroke; quality of life; walking speed
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic group (Experimental): This group receives conventional rehabilitation plus robotic exoskeleton-assisted gait rehabilitation.
  Interventions: Device: Robotic exoskeleton-assisted gait rehabilitation
- Control group (Active Comparator): This group receives conventional rehabilitation alone.
  Interventions: Other: Conventional rehabilitation

INTERVENTIONS:
Device: Robotic exoskeleton-assisted gait rehabilitation — Use a robotic exoskeleton for gait rehabilitation in addition to conventional rehabilitation
  Arms: Robotic group
Other: Conventional rehabilitation — Regular post-stroke rehabilitation
  Arms: Control group

SUMMARY:
Investigators aimed to examine the effectiveness of robotic exoskeleton-assisted gait training in stroke rehabilitation, and to determine predicting factors of significant improvements in post-stroke patients. Investigators hypothesized that robotic assisted gait training brings better strength recovery and functional improvement.

ELIGIBILITY:
Inclusion Criteria:

* patients aged from 30 to 80 years
* hemiparesis due to ischemic or hemorrhagic stroke in the last 6 months

Exclusion Criteria:

* with a significant history of pain or injury of lower limbs that affected their walking ability,
* with cardiopulmonary diseases that prohibited exercise training
* with impaired cognitive function
* unable to complete the timed up-and-go test
* able to complete the timed up-and-go test in <20 seconds using walking device

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline distance walked in 6 minute walk test after entire rehabilitation program (4 weeks) | 4 weeks
Change from baseline time needed to complete Timed-Up-and-Go test after entire rehabilitation program (4 weeks) | 4 weeks
Change from baseline scores in 12-item short form survey after entire rehabilitation program (4 weeks) | 4 weeks
  12-item short form survey (SF-12): scores range from 0 to 100, with higher scores indicating better physical and mental health functioning
Change from baseline Isokinetic strength after entire rehabilitation program (4 weeks) | 4 weeks
  tested by isokinetic dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No